CLINICAL TRIAL: NCT04107480
Title: PRolaCT - Three Multicenter Prolactinoma Randomized Clinical Trials
Brief Title: PRolaCT - Three Prolactinoma RCTs
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, I.M. Zandbergen, MD, Coordinating Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRolaCT; 843002806 (Other Grant/Funding Number: ZonMw); NL63919.058.18 (Registry Identifier: CCMO-registry)
Record Dates: First submitted 2019-08-27; First posted 2019-09-27 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Prolactinoma; Prolactin-Producing Pituitary Tumor
Keywords: prolactinoma; dopamine agonist; endoscopic trans-sphenoidal adenoma resection; remission rate; health-related quality of life
MeSH Terms: conditions — Prolactinoma | interventions — Dopamine Agonists; Standard of Care

STUDY DESIGN:
Intervention Model Description: This partially randomized, preference trial design, comprises three unblinded randomized controlled trials (RCTs) and an observational study arm (PRolaCT-O) that compare neurosurgical counselling and potentially subsequent endoscopic transsphenoidal adenoma resection with current standard care (DA treatment). Patients with a non-invasive prolactinoma of limited size (<2.5 cm) will be divided over the three RCTs based on duration of pre-treatment with DA: PRolaCT-1: newly diagnosed, treatment naive patients; PRolaCT-2: patients with limited duration of DA treatment (4-6 months); and PRolaCT-3: patients with persisting prolactinoma after DA treatment for >2 years. PRolaCT-O will include patients who decline randomization or those with a clear treatment preference. After study inclusion and treatment allocation, all study procedures and follow up are equal for the three RCTs and PRolaCT-O and are therefore discussed as one.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in the intervention groups will be referred to one of the participating neurosurgical centers, for surgical consultation. After this consultation, the patient may choose to continue with surgery or not.
  Interventions: Procedure: Endoscopic trans-sphenoidal adenoma resection
- Standard care (Active Comparator): Patients in the standard care groups will receive treatment as usual as described by the US Endocrine Society.
  Interventions: Drug: Dopamine Agonists

INTERVENTIONS:
Procedure: Endoscopic trans-sphenoidal adenoma resection — Neurosurgical consultation consists of at least one consult with a neurosurgeon and at least one consult with an endocrinologist with relevant experience. If the multidisciplinary team (MDT) agrees the patient is a good surgical candidate, the patient is asked consent for surgery, as is a custom part of preoperative requirements. When the patient decides not to have the surgery, (s)he will receive standard medical treatment, but will continue study follow up in the intervention group.
  Surgery only takes place if both the MDT and the patient agree to it and should then be planned within three months after randomization. Surgery is performed by one or two trained neurosurgeons in the hospital where the counseling took place. A standard, semi-protocolled, endoscopic trans-sphenoidal surgical resection of the prolactinoma is performed according to standard practice.
  Arms: Intervention
Drug: Dopamine Agonists — The treating physician adheres to the treatment protocol in general, but has freedom to choose treatment to his/her ideas how to deliver best care.
  Current first line treatment consists of a dopamine agonists: cabergoline (currently the most used), bromocriptine or quinagolide. All dopamine agonists are taken orally, and the dosage may be raised based on its effect. It is usually titrated to achieve a normal or suppressed prolactin level and restoration of the gonadal axis. Dopamine agonist treatment is discontinued after 2 years of treatment, unless a normal prolactin level cannot be achieved. The dopamine agonist is restarted when prolactin levels rise after the medication is discontinued.
  In standard care, surgical treatment is reserved for patients who don't tolerate medication, or whose adenoma fails to show a sufficient response. Patients in the control group with an intolerance for dopamine agonists or an insufficient response may be offered surgery as part of standard care.
  Other Names: Standard Care
  Arms: Standard care

SUMMARY:
This study aims to investigate if endoscopic trans-sphenoidal prolactinoma resection as a first line treatment, or as an equally valid second line treatment after a short (4-6 months) or long (>2 years) period of pretreatment with a dopamine agonist is superior to standard care for several outcome parameters. The main objectives are to investigate this for quality of life and remission rate. The secondary objectives are to investigate this for biochemical disease control, recurrence rates, clinical symptom control, tumor shrinkage on MRI, pituitary functioning, the occurrence of adverse reactions to treatment, disease burden, and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* A history of signs and symptoms compatible with the diagnosis prolactinoma.
* New, recent (PRolaCT-1) or known diagnosis of hyperprolactinaemia, defined as a prolactin level 2 times the local laboratory maximum. At the time of randomization hyperprolactinaemia is still present, or was present < 12 months before inclusion (PRolaCT-2 and PRolaCT-3).
* No clear alternative explanation for hyperprolactinaemia, e.g. medication use.
* Presence of a clearly identifiable (persisting) pituitary mass on MRI not invading the cavernous sinus and having an optimal chance to be completely resected (generally adenomas with a maximum diameter nog exceeding 25mm). A representative MRI at the time of randomization is required, this MRI should generally not be older than 12 months in PRolaCT-3 and 2 months in PRolaCT-1 and PRolaCT-2.
* Competent and able to fill in questionnaires.
* One of the following, dividing patients in to our three RCTs:

  * PRolaCT-1: no prior treatment for prolactinoma;
  * PRolaCT-2: treatment with a dopamine agonist for 4-6 months; or
  * PRolaCT-3: treatment with a dopamine agonist for at least 2 years.

Exclusion Criteria:

* Contraindication for one of the treatment modalities, e.g. severe side effect of cabergoline, contraindications to surgery, or a clear indication for surgical resection.
* Pregnancy at the time of randomization.
* Clinical acromegaly.
* Prior pituitary gland surgery or radiotherapy to the pituitary gland area.
* Severe renal failure (eGFR <30 ml/min).
* Insufficient understanding of the Dutch or English language.
* Other medical conditions that to the opinion of the physician are not compatible with inclusion in a trial.

Patients eligible for participation in one of the RCTs, but do not consent to randomisation or in whom there is a clear patient or physician preference for either DA treatment or surgery, are considered for participation in PRolaCT-O.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life | 12 months after randomization/baseline
  Health-Related Quality of Life is defined as the score on the mental health scale of the Medical Outcomes Study (MOS) Short-Form Health Survey (SF-36), measured at T=12.
Long-term remission | 36 months after randomization/baseline
  Disease remission is defined as normoprolactinaemia (a prolactin level below the upper limit of normal as defined by the laboratory site where it is measured), in the absence of dopamine agonist treatment for at least 3 months or an actual pregnancy that was established during at least 3 months absence of dopamine agonist treatment, measured at T=36.

SECONDARY OUTCOMES:
Short-term remission | 27 months after randomization/baseline
  Disease remission as defined under the primary outcome for remission, measured at T=27.
Very long-term remission | 60 months after randomization/baseline
  Disease remission as defined under the primary outcome for remission, measured at T=60
Biochemical disease control | 12 months after randomization/baseline
  Biochemical disease control is defined as normoprolactinaemia (a prolactin level below the upper limit of normal as defined by the laboratory site where it is measured), or an actual pregnancy, with or without the use of a dopamine agonist, measured at T=12.
Recurrence rate | 36 and 60 months after randomization/baseline
  Disease recurrence is defined as recurrence of hyperprolactinaemia (a prolactin level >2 times the upper limit of normal as defined by the laboratory site where it is measured) in the absence of dopamine agonist treatment, after a period of normoprolactinaemia (without dopamine agonist treatment). This is measured only in patients who have achieved disease remission at T=27, and is measured at T=36 and T=60.
Clinical symptom control | 12, 27, 36 and 60 months after randomization/baseline
  Clinical symptom control is defined as the absence of physical and psychiatric symptoms of prolactinoma.
Tumor shrinkage on MRI | 12 and 36 months after randomization/baseline
  Tumor growth or shrinkage will be calculated as the percentage difference from baseline in tumor size (defined as the maximal diameter measured in mm) and tumor volume (calculated using Cavalieri's principle: tumor volume = 4/3 × pi (a/2 × b/2 × c/2) where a, b and c represent the diameters (in mm) in the 3 dimensions), measured at T=12 and T=36. It will be considered as a relevant shrinkage if tumor diameter or volume decreases at least 20%.
Pituitary functioning | 12 and 36 months after randomization/baseline
  The functioning of the pituitary axes other than prolactin (i.e. gonadal, thyroidal, corticoid, growth hormone and ADH axes), measured when indicated upon judgement by the treating physician (e.g. when an axis was deviant at baseline of as part of routine follow up after surgery) at T=12 and T=36.
  A pituitary axis will be considered normal when the associated measurement is within its normal range specific to the laboratory where it was measured in the absence of supplement treatment.
Complications | Baseline and 12 months after randomization/baseline
  Treatment specific adverse effects:
  - The occurrence of known complications to surgery (i.e. cerebrospinal fluid leakage, diabetes insipidus, syndrome of inappropriate ADH-secretion, nasal complaints, decreased sense of smell/taste, intradural hemorrhage, meningitis, visual loss or a new pituitary deficit), as documented in patients' medical records by the treating physician, measured at T=12.
Side effects | Baseline and 12, 27 and 36 months after randomization/baseline
  Treatment specific adverse effects:
  - Occurrence of known side effects to dopamine agonist treatment as documented with the National Cancer Institute Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE™) and a combined Impulse Control Disorder questionnaire at baseline, T=12, T=27 and T=36.
Health-Related Quality of Life | Baseline and 12, 27, 36 and 60 months after randomization/baseline
  Described by the scores on all sub-scales of the SF-36, in addition to the primary outcome on health-related quality of life. Measured at baseline, T=12, T=27, T=36 and T=60.
Depression and anxiety scores | baseline and 12 and 36 months after randomization/baseline
  Measured with the Hospital Anxiety and Depression Scale (HADS). This questionnaire uses 14 items; seven related to anxiety and seven to depression, to calculate anxiety and depression scores, ranging from 0 to 21.
Disease burden | baseline and 12, 36 and 60 months after randomization/baseline
  Measured with the Leiden Bother and Needs Questionnaire at baseline, T=12, T=36 and T=60.
Healthcare costs | Every 6 months until 36 months after randomization/baseline
  Measured every 6 months until T=36, with the iMTA Medical Consumption Questionnaire.
Non-healthcare costs | Every 6 months until 36 months after randomization/baseline
  Measured every 6 months until T=36, with the iMTA Productivity Cost Questionnaire.
Quality-Adjusted Life Years (QALYs) | Baseline and 6, 9, 12, 18, 24, 27, 30 and 36 months after randomization/baseline
  Measured at 3-6 month intervals, with the EQ-5D-5L.

CONTACTS AND LOCATIONS:
Overall Officials: Nienke R Biermasz, MD, prof., Principal Investigator — Endocrinologist LUMC; Wouter R van Furth, MD, PhD, Principal Investigator — Neurosurgeon LUMC
Locations (3):
- Netherlands (3):
  - Amsterdam University Medical Center, loc. AMC, Amsterdam-Zuidoost, North Holland
  - Reinier de Graaf Gasthuis, Delft, South Holland
  - Leiden University Medical Center, Leiden, South Holland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zandbergen IM, Zamanipoor Najafabadi AH, Pelsma ICM, van den Akker-van Marle ME, Bisschop PHLT, Boogaarts HDJ, van Bon AC, Burhani B, le Cessie S, Dekkers OM, Drent ML, Feelders RA, de Graaf JP, Hoogmoed J, Kapiteijn KK, van der Klauw MM, Nieuwlaat WCM, Pereira AM, Stades AME, van de Ven AC, Wakelkamp IMMJ, van Furth WR, Biermasz NR; Dutch Prolactinoma Study Group. The PRolaCT studies - a study protocol for a combined randomised clinical trial and observational cohort study design in prolactinoma. Trials. 2021 Sep 25;22(1):653. doi: 10.1186/s13063-021-05604-y. PMID 34563236